CLINICAL TRIAL: NCT05098795
Title: Training Peer Recovery Coaches to Promote Retention and Adherence to Medications for Opioid Use Disorder Among Low-Income Adults
Brief Title: FOREward Together: Training Peer Recovery Coaches to Promote Retention and Adherence to MOUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Julia Felton, Assistant Scientist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEP: 14920-29
Record Dates: First submitted 2021-10-07; First posted 2021-10-28 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use
Keywords: Medications for opioid use disorder; Peer recovery coach; Substance use; Behavioral activation; Task sharing; Treatment retention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-delivered Behavioral Activation (Experimental): Adults 18 years or older on MOUD or referred to MOUD will receive Behavioral Activation (BA) an evidence-based intervention (EBI) by trained Peer Recovery Coaches (PRC)
  Interventions: Behavioral: Behavioral Activation (BA)

INTERVENTIONS:
Behavioral: Behavioral Activation (BA) — BA seeks to increase the positive reinforcement patients experience from their natural environment by promoting prosocial and valued experiences. BA has been found to improve substance use treatment retention and adherence, as well as medication adherence in low-income individuals with HIV/AIDS.

SUMMARY:
This project aims to implement a peer-led intervention to support retention and adherence to medications for opioid use disorder among low-income adults in Detroit, as well as a training manual for peer recovery coaches serving similar populations. The approach will serve as a guide to coaches in providing positive reinforcement and helping those in treatment to schedule and engage in valued activities. Researchers will examine the effectiveness of the intervention, supervision and training models, and share results with policymakers and treatment programs.

DETAILED DESCRIPTION:
Low-income and racial/ethnic minorities suffer disproportionately from the opioid use disorder (OUD) crisis, evidencing consistently lower rates of critical treatment outcomes, including medication for OUD (MOUD) engagement and retention. While these individuals exhibited a need for evidence-based care prior to the pandemic, low-income, racial/ethnic minority populations have been disproportionately affected by COVID-19, as have persons with SUDs.

Peer Recovery Coaches (PRC) are individuals with lived-experiences with substance use who have been certified by the state to assist in treatment recovery. Because of similarities between PRCs and substance use clients, PRCs can overcome many of the barriers that clients face to engaging and staying in MOUD treatment, such as stigma. goal of the current project is to conduct an open-label pilot trial to examine the feasibility, acceptability and accessibility of a PRC-led intervention to support retention in MOUD care.

This project proposes to develop a novel and sustainable model for improving retention in MOUD treatment by training PRCs to deliver an evidence-based intervention (EBI), Behavioral Activation (BA). BA seeks to increase the positive reinforcement patients experience from their natural environment by promoting prosocial and valued experiences. BA has been found to improve substance use treatment retention and adherence, as well as medication adherence in low-income individuals with HIV/AIDS. To that end, the following goal is proposed: to evaluate the preliminary feasibility, acceptability, and effectiveness of the PRC- delivered BA approach. An open-label pilot trial (n=40) of the adapted PRC-delivered BA intervention and training protocol in a representative agency in Detroit, MI serving a low-income, predominantly African-American population will be conducted. Findings from this phase of the project will be used to re-adapt the manual and training procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participants must (1) be receiving or referred to MOUD; and (2) be over the age of 18.

Exclusion Criteria:

* Exclusion criteria will be (1) demonstrating active, unstable or untreated psychiatric symptoms, including mania and/or psychosis; or (2) inability to understand the study and give informed consent in English Active, Unstable or Untreated Psychiatric Symptoms: The study team is committed to recruiting a sample that reflects the complexity and likely comorbidity of people with moderate to severe OUD in this setting. Therefore, only people whose concurrent mental health issues preclude ability to participate with the procedures in this study will be excluded. Throughout the study, researchers will monitor for active, unstable or untreated psychiatric symptoms as the presence of these symptoms during study procedures would interfere with participation. Monitoring for exclusionary psychiatric symptoms can include reviewing data in medical chart (per protocol-approved access to medical records), observation during assessments and intervention sessions, and/or current symptoms detected on the MINI modules for psychosis and mania.

Inability to complete informed consent/ study in English. This study/intervention will be implemented in English only. Therefore, the capacity and willingness to give written informed consent in English, to understand the study and inclusion and exclusion criteria in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Felton, PhD., Principal Investigator — Henry Ford Health System
Locations (1):
- The Detroit Recovery Project, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
After all primary analyses are complete, de-identified data will be available per request of outside individual

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled via flyers and word-of-mouth at a community-based substance use treatment setting from December 2021 through April 2023.
Period: Overall Study
Arm/Group | Peer-delivered Behavioral Activation
Started | 29
Started BA (Engaged in at least one Behavioral Activation session) | 21
Completed BA (Completed the BA intervention, defined as taking part in at least 8 sessions.) | 13
Completed Post-assessment (Completed follow-up (post) assessment measures) | 12
Completed | 12
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Peer-delivered Behavioral Activation
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: MOUD Retention Rate
Description: Average number of days a participant missed an MOUD appointment between receiving the intervention and completing the follow-up assessment (approximately 8-12 weeks following the intervention date), averaged across all participants with available data.
Time Frame: Measured between participants' completion of baseline assessment and completion of the follow-up assessment (approximately 8-12 weeks following the intervention date).
Population: We were able to get data on MOUD visits from 18 participants from the total sample.
Measure: Mean (Standard Deviation); unit: number of days missed MOUD appointment
Arm/Group | Peer-delivered Behavioral Activation
Number analyzed (Participants) | 18
number of days missed MOUD appointment | .42 (2.86)

2. Primary Outcome: Intervention Fidelity: Proportion of Intervention Components Delivered as Intended
Description: Defined as the proportion of all 24 intervention components in the total intervention that were delivered with fidelity by the interventionist (ranging from 0 to 1.0 with higher proportion reflecting more fidelity).
Time Frame: The number of days between starting the intervention and completing the intervention (approximately 8-10 weeks).
Population: Fidelity was examined among participants who took part in at least one BA session.
Measure: Mean (Standard Deviation); unit: proportion of elements delivered
Arm/Group | Peer-delivered Behavioral Activation
Number analyzed (Participants) | 21
proportion of elements delivered | .83 (.09)

3. Secondary Outcome: Intervention Acceptability: Percentage of Patients Enrolled Who Attend ≥75% Sessions
Description: Defined as the percentage of participants who started the intervention who then finish the intervention (defined as completing 8 total sessions)
Time Frame: The number of days between starting the intervention and completing the intervention (approximately 8-10 weeks).
Population: We examined the percentage of all participants who started the intervention who then completed the intervention (defined as taking part in 8 sessions)
Measure: Number; unit: percentage of participants
Arm/Group | Peer-delivered Behavioral Activation
Number analyzed (Participants) | 21
percentage of participants | 62

4. Secondary Outcome: Intervention Feasibility: Percentage of Patients Who Consents Who Started BA
Description: Defined as the percentage of participants who started BA sessions relative to those who enrolled in the program
Time Frame: The number of days between starting providing consent and starting BA (approximately 1-5 weeks).
Population: We examined the percentage of participants who took part in at least one BA session relative to those who enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer-delivered Behavioral Activation
Number analyzed (Participants) | 29
Participants | 21

ADVERSE EVENTS:
Time Frame: Over the course of the intervention delivery, approximately one year.
Description: No differences in how adverse events are described
Arm/Group | Peer-delivered Behavioral Activation
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
None noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT05098795/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/95/NCT05098795/SAP_001.pdf